CLINICAL TRIAL: NCT04158453
Title: A Randomised, Double-blind, Placebo-controlled, Single and Repeated Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AUT00201 in Healthy Male and Female Volunteers
Brief Title: Safety, Blood Levels and Effects of AUT00201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autifony Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUT011201
Record Dates: First submitted 2019-11-07; First posted 2019-11-08 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AUT00201 (Active Comparator)
  Interventions: Drug: AUT00201
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AUT00201 — Oral dose of AUT00201
  Arms: AUT00201
Drug: Placebo — Oral dose of placebo
  Arms: Placebo

SUMMARY:
The study medicine is a potential future treatment for schizophrenia, an illness that affects the way that people think, feel or behave. It is not clear what causes schizophrenia, but it's been linked to chemical imbalance in the brain. It is hoped that the study medicine will activate specific sites in the brain to help correct that imbalance. Current treatments for schizophrenia don't work very well and can cause unpleasant side effects. It is hoped that the study medicine will work better, and have fewer side effects than existing medicines.

In this 2 part study (Part A: up to 40 healthy male subjects and up to 8 healthy female subjects, Part B: up to 32 healthy male subjects) the primary aim is to assess how safe the study medicine is in healthy men and women.

This study will be in 2 parts, as follows:

Part A will assess single doses of AUT00201 and Part B will assess multiple doses. Part A will be divided into 3 sub-parts: Part A1 will assess single ascending doses in healthy men, Part A2 will assess single ascending doses in healthy women, and Part A3 will assess the effect of food on the PK of AUT00201 in healthy men.

A pharmaceutical company, Autifony Therapeutics Limited, is funding the study. The study will take place at 1 centre in London.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive male (all groups except Part A2) or female (Part A2 only) volunteers
* Must have body mass index (BMI) of 18.0-31.0 kg/m2
* Must be healthy based on clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine
* Must be able to give fully informed written consent.

Exclusion Criteria:

History or presence of

* Epilepsy
* Severe head injury, or any other chronic neurological condition or any psychiatric disorder
* Abnormal screening EEG (Part A1 and Part B only)
* Positive tests for hepatitis B & C, HIV
* Severe adverse reaction to any drug
* Sensitivity to trial medication
* Drug or alcohol abuse
* Use of over-the-counter medication within previous 7 days (with the exception of Paracetamol [acetaminophen])
* Prescribed medication during previous 28 days
* Participation in other clinical trials of unlicensed medicines
* Loss of more than 400 mL blood, within the previous 3 months
* Vital signs or QTcF interval outside the acceptable range
* Clinically relevant abnormal findings at the screening assessment
* Acute or chronic illness
* Clinically relevant abnormal medical history or concurrent medical condition
* Positive result for suicidal ideation or behaviour using the Colombia suicide severity rating scale (C-SSRS)
* Possibility that volunteer will not cooperate
* Pre-menopausal females who are pregnant or lactating, or who are sexually active and not using a reliable method of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with treatment-related adverse events | Study Duration (2 weeks post last dose)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No